CLINICAL TRIAL: NCT04656600
Title: A Single Arm, Prospective, Open Label, Multicenter Study to Evaluate Efficacy and Safety of One-year Maximum Dosage in Chinese Label of Imiglucerase Treatment in Chinese Patients Who Are Diagnosed as Gaucher Disease Type Ⅲ
Brief Title: Study to Evaluate Efficacy and Safety of Imiglucerase Treatment in Chinese Patients With Gaucher Disease Type Ⅲ
Acronym: SEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16031; U1111-1244-1166 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Gaucher's Disease
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerezyme® / Imiglucerase (Experimental): Cerezyme® (imiglucerase for injection) is administered by intravenous infusion, 60 U/kg once every 2 weeks.
  Interventions: Drug: Cerezyme® / Imiglucerase

INTERVENTIONS:
Drug: Cerezyme® / Imiglucerase — Pharmaceutical form: lyophilisate for solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective

* To evaluate the efficacy on hematologic manifestations of imiglucerase treatment in Chinese patients who are diagnosed as Gaucher disease type Ⅲ
* To evaluate the safety profile of imiglucerase in maximum dose in the label (60U/kg, IV biweekly) in Chinese patients.

Secondary Objective

* To evaluate the efficacy on viscera manifestations of imiglucerase treatment in Chinese patients who are diagnosed as Gaucher disease type Ⅲ
* To evaluate the efficacy on bone disease of imiglucerase treatment in Chinese patients who are diagnosed as Gaucher disease type Ⅲ
* To evaluate the effect on quality of life of imiglucerase treatment in Chinese patients who are diagnosed as Gaucher disease type Ⅲ

DETAILED DESCRIPTION:
Approximatively 14 months including a 12 months treatment period

ELIGIBILITY:
Inclusion criteria:

* Capable of giving signed informed consent.
* Participant is diagnosed with GD type Ⅲ
* Participant with neurological manifestations
* Participant whose age is > 2 years old.
* Participant whose spleen and/or liver volume is > ULN at Screening.

Exclusion criteria:

* Major congenital anomaly
* Clinically significant intercurrent organic disease unrelated to Gaucher disease, which means the disease or condition that may have impact on the parameters chosen for primary endpoints (e.g. level of hemoglobin platelets, liver/spleen enlargement and bone pains)
* Prior treatment with ERT.
* Physical conditions that cannot tolerate regular treatment or follow-up visit.
* Pregnant or lactating women
* Participant is participating in or has participated in another clinical study using any investigational therapy in 3 months
* Participant has been diagnosed with central nervous system disease unrelated to Gaucher disease, or MRI result of the participant indicates space-occupying lesion in central nervous system
* The patient has a documented hemoglobinopathies, deficiency of iron, vitamin B-12, or folate that requires treatment not yet initiated or, if initiated, the patient has not been stable under treatment for at least 6 months prior to administration of the first dose of Cerezyme in this study
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Any specific situation during study implementation/course that may rise ethics considerations
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Changes in haemoglobin | Baseline to the end of 12 months
  The mean changes in haemoglobin
Changes in platelet count | Baseline to the end of 12 months
  The mean changes in platelet count
Adverse events | Baseline to the end of 13 months
  Number of participants with AEs

SECONDARY OUTCOMES:
Changes in spleen volume | Baseline to the end of 12 months
  The mean change of spleen volumne
Changes in liver volume | Baseline to the end of 12 months
  The mean change of liver volumne
Skeletal involvement | Baseline to the end of 12 months
  The changes in frequency, duration and severity of bone pain and number of bone crisis The changes in frequency, duration and severity of bone pain and number of bone crisisThe changes in frequency, duration and severity of bone pain and number of bone crisis
Quality of life (QoL) | Baseline to the end of 3 months, 6 months, 9 months and 12 months
  The mean change of QoL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- China (5):
  - Investigational Site Number : 107, Beijing
  - Investigational Site Number : 101, Beijing
  - Investigational Site Number : 104, Chengdu
  - Investigational Site Number : 102, Guangzhou
  - Investigational Site Number : 105, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16031 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25278&tenant=MT_SNY_9011